CLINICAL TRIAL: NCT07301554
Title: Evaluation of Food Preferences in Patients Treated Surgically for Craniopharyngiomas
Brief Title: Food Preferences and Craniopharyngiomas
Acronym: PREFAMHYPO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250745; 2025-A02014-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Craniopharyngioma
Keywords: Craniopharyngioma; food preferences; changes
MeSH Terms: conditions — Craniopharyngioma; Food Preferences

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- groups 1: Craniopharyngioma patients: 40 adults surgically treated for craniopharyngioma (≥ 3 months post-surgery).
- Control participants: 80 adults without hypothalamic-pituitary disease, matched on age, sex, and BMI with groups 1 and 2.
- groups 2: Pituitary macroadenoma patients: 40 adults surgically treated for pituitary macroadenoma with ≥ 2 anterior pituitary hormone deficiencies.

SUMMARY:
The hypothalamus plays a key role in regulating appetite, satiety, and energy balance. When tumors such as craniopharyngiomas develop in this region, they can disrupt these mechanisms and lead to a form of severe weight gain known as hypothalamic obesity. Several factors play a role in the development of hypothalamic obesity that is often resistant to traditional treatments. Changes in food preferences notably a higher liking for food rich in fat and sugar may be implicated as has been reported in common obesity.

The working hypothesis of the study is that hypothalamic lesions may alter food preferences, leading to an increased preference for high-fat and high-sugar foods, and that these changes in dietary choices contribute among other factors to the development of hypothalamic obesity.

By providing the first evaluation of food preferences in adults treated surgically for craniopharyngiomas, this study will shed light on the role of hypothalamic lesions in modifying dietary choices. The results may help explain why some patients experience rapid and resistant weight gain, and could guide future strategies to better manage hypothalamic obesity.

DETAILED DESCRIPTION:
Hypothalamic obesity is a rare but severe condition characterized by rapid and often refractory weight gain following hypothalamic lesions. Among suprasellar tumors, craniopharyngiomas are the most frequent, and up to 40% of patients present with obesity at diagnosis. Over the course of treatment, including surgical management, the prevalence of obesity may rise to 60%. The most pronounced weight gain typically occurs within the first year after surgery. This weight increase is multifactorial, involving hypothalamic damage to nuclei regulating appetite and satiety, neuroendocrine dysfunction, reduced basal metabolic rate, decreased physical activity, and autonomic imbalance leading to hyperinsulinism. Additional contributors include neurocognitive and sleep disturbances, visual impairment, and medication side effects.

Beyond the quantitative increase in food intake, food palatability is a key determinant of dietary choices and caloric intake. Highly palatable foods, generally rich in fats and sugars, stimulate brain reward circuits, reinforcing their consumption and thereby promoting excess caloric intake and weight gain. While such mechanisms have been described in common obesity, food preferences have never been systematically investigated in patients with hypothalamic lesions, particularly those with craniopharyngiomas. Animal studies suggest that the lateral hypothalamus plays a critical role in responses to addictive substances as well as to fat and sugar consumption, raising the hypothesis that hypothalamic tumors may alter food preferences in humans and contribute to hypothalamic obesity.

This study, entitled PREFAMHYPO, is a two-phase, non-interventional observational clinical investigation designed to explore the role of food preferences in hypothalamic obesity.

Study Objectives and Design

The study has two main phases:

The objective of Phase 1 is the cultural adaptation and psychometric validation of the French version of the Food Preference Questionnaire (FPQ). The questionnaire, which assesses preferences across major food categories, has been translated and back-translated to ensure accuracy. This phase will confirm its reliability and validity in a French adult population, using measures such as internal consistency (Cronbach's alpha), test-retest reproducibility, and exploratory factor analysis. A subgroup of 50 participants will complete the FPQ twice, two weeks apart, to assess reproducibility.

Phase 2 consists of a cross-sectional evaluation of food preferences using the validated FPQ in three groups :

* Adults surgically treated for craniopharyngiomas
* Adults surgically treated for pituitary macroadenomas with at least two anterior pituitary hormonal deficits matched to craniopharyngioma patients on age, sex, and body mass index (BMI).
* Control participants without hypothalamic-pituitary disease matched to craniopharyngioma patients on age, sex, and body mass index (BMI).

The primary objective of this second phase is to compare food preferences across groups, with a specific focus on preferences of high-fat and high-sugar foods. Secondary objectives include evaluation of fat preferences, evaluation of eating behavior via the validated French version of DEBQ, evaluation of physical activity via the validated version of IPAQ, anthropometrics, body composition, and standard hormonal/metabolic panels.

Study Procedures

For phase 1, after receiving detailed information and providing documented non-opposition, participants will complete a set of standardized, self-administered questionnaires at inclusion and only 50 participants will complete the questionnaires again after 14 days.

For phase 2, after receiving detailed information and providing documented non-opposition, participants will complete a set of standardized, self-administered questionnaires at inclusion during a routine consultation or hospitalization, with no subsequent follow-up.

For patients, relevant anthropometric, clinical, and biological data will be retrieved from medical records, including BMI, waist circumference, hormone levels, metabolic parameters, treatments, comorbidities, and surgical details.

Data Management and Quality Assurance

Data will be collected by investigators at participating AP-HP sites and entered into a secure, password-protected REDCap system or encrypted Excel database. Patient anonymity will be preserved through pseudonymization, using site codes, inclusion numbers, and initials. The link between codes and identities will be kept locally under investigator control.

Source documents include medical records, consultation reports, surgical notes, laboratory results, imaging reports, and the completed questionnaires. All gathered data relevant to this study will be retained for 15 years, in accordance with French regulations. Only authorized study personnel or monitors will have access, under conditions ensuring confidentiality and compliance with Good Clinical Practice (GCP).

Data quality will be ensured through predefined validation rules, consistency checks, and central monitoring by the sponsor (AP-HP). Statistical analyses will be performed on pseudonymized datasets.

Sample Size and Statistical Analysis

The sample size for Phase 1 is based on Cattell's method, requiring at least three participants per item. With 62 FPQ items, 186 participants are needed.

For Phase 2, the rarity of craniopharyngiomas necessitates an exploratory design with 40 cases, 40 macroadenoma patients, and 80 controls. This sample is sufficient to provide descriptive and comparative analyses, generate hypotheses, and inform future larger-scale studies.

Statistical methods include

Phase 1 : Exploratory factor analysis (principal component analysis with Varimax rotation), Cronbach's alpha for internal consistency, intraclass correlation coefficients for reproducibility, and validity testing against external constructs (e.g., psychological distress measured by Kessler-10).

Phase 2 : Descriptive statistics, ANOVA or Kruskal-Wallis tests for group comparisons, post hoc multiple comparison tests, correlation analyses (Pearson or Spearman), and multivariable linear regression models to identify independent factors associated with food preferences. Missing data will be handled using appropriate statistical techniques, including imputation when necessary.

Duration

The total study duration is estimated at 36 months, including 24 months of participant recruitment and 12 months for data analysis and reporting.

Inclusion of participants for Phase 1 will be done within three months and for phase 2 within 21 months. Each participant's involvement is limited to one visit except for the Phase 1 subgroup completing the retest at 14 days.

Ethical Considerations

This is a non-interventional observational study with minimal risk. No experimental treatments or invasive procedures are involved. All participants will be informed orally and in writing, and their non-opposition to participation will be documented before any data collection. The study complies with French regulations governing research involving human participants, data protection (GDPR), and Good Clinical Practice.

The sponsor of the study is Assistance Publique - Hôpitaux de Paris (AP-HP), with coordination by the Endocrinology, Diabetology and Nutrition Department at Ambroise Paré Hospital, and collaboration with the Neurosurgery Department at Lariboisière Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criteria: complete medical record accessible, capacity to understand and complete self-administered questionnaires, agreement to complete the questionnaires at the time of inclusion, adult subject, not in an emergency situation, provision of non-opposition (opt-out consent documented), affiliation to a social security scheme.

Inclusion (Phase 1): Adults residing in France, aged 18 - 74 years from the general population.

Inclusion (Phase 2): Adults aged 18 - 74 years;

Group 1: patients with craniopharyngioma surgery ≥ 3 months prior to inclusion.

Group 2: patients with pituitary macroadenoma surgery with documented ≥ 2 anterior pituitary deficits.

Group 3: Follow-up for an endocrine condition without hypothalamo-hypophyseal involvement, acceptable conditions (thyroid nodule without dysthyroidism, PCOS, peripheral hirsutism, calcium metabolism disorders), no known treatments or prior medical history likely to influence eating behaviour.

Exclusion Criteria:

* Common exclusion criteria: bariatric surgery, GLP-1 agonist treatment, chronic disease affecting alimentation, pregnancy or breastfeeding, specific diets (gluten-free, vegetarian, vegan...), refusal or opposition to data use, vulnerability status (under guardianship or legal protection) or inability to complete questionnaires or to understand the proposed research or to express a clear opinion regarding non-opposition.

Additional exclusion criteria:

phase 1: Type 1 or type 2 diabetes, Active smoking, alcohol misuse, drug use, diagnosed psychiatric disorders or eating behaviour disorders.

Phase 2:

Person benefiting from State Medical Aid (AME).

Control group:

Hypothalamo-hypophyseal pathology, type 1 or type 2 diabetes, uncontrolled hyperthyroidism or hypothyroidism, adrenal hormone hypersecretion disorder, history of or ongoing treatment for active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1 : Adult French residents aged 18 - 74 years from the general population (n=186) for FPQ validation (recruited among hospital staff, patients, accompanying persons).
  Phase 2 : Adults aged 18 - 74 years in three groups (40 patients with craniopharyngiomas, 40 matched patients with macroadenomas with ≥2 hormonal deficits , 80 matched controls); total n=160 for phase 2.
  Overall total across phases = 346 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Psychometric validation of the French food preference questionnaire (FPQ): phase 1 | at baseline
  Validation of the French version of the Food Preference Questionnaire (FPQ) in an adult population in France. The Food Preference Questionnaire (FPQ) is the primary tool used to evaluate participants' food preferences for 62 food items, such as meats, dairy products, cereals, fruits, vegetables, and snack foods. For each item, participants indicate their degree of liking using a 6-point response scale from "dislike strongly" to "like strongly" ("Do not like at all", "Dislike moderately", "Neutral", "Like a little", "Like very much", "Not applicable"), allowing quantification of preference intensity across food types.
  Validity will be evaluated through exploratory and confirmatory factor analyses, while reliability will be assessed using internal consistency (Cronbach's alpha coefficient) and reproducibility (test-retest).
Evaluation of scores measuring FPQ: phase 2 | at baseline
  The main objective is to characterize food preferences in patients operated on for a craniopharyngioma by comparing them with two control groups: patients operated on for a pituitary macroadenoma with anterior pituitary insufficiency, and a control population matched for age, sex, and body mass index (BMI), calculated as mass (kg) /(height in m)^2. The questionnaire validated in phase 1 will be used and questionnaire results will be analyzed quantitatively to identify specific food preference profiles within each group and to explore potential associations with clinical and metabolic parameters.

SECONDARY OUTCOMES:
Evaluation of the Fat Preference | at baseline
  Phase 2 :
  Evaluation of the liking and consumption frequency between higher-fat and lower-fat versions of common foods (e.g., baked potato versus French fries, full-fat versus reduced-fat ice cream).
  It uses forced-choice items with three components per food pair : "have you eaten this food?", "which tastes better?", and "which do you eat most often?".
Evaluate of eating behaviors | at baseline
  Phase 2 :
  Tool: Dutch Eating Behavior Questionnaire (DEBQ). Assessment of eating behaviors (emotional, restrained, external). The DEBQ has been translated and validated in 14 languages, including French. Each item uses a 5-point scale ("Never", "Rarely", "Sometimes", "Often", "Very often"). Higher scores indicate higher levels of the corresponding eating behavior.
Assessment of physical activity | at baseline
  Phase 2:
  Tool: International Physical Activity Questionnaire (IPAQ) Measurement of physical activity level over the previous 7 days. Higher scores reflect higher physical activity levels. It has been validated in several languages, including French.
Collecte of BMI | at baseline
  Body Mass Index (BMI): BMI = (weight (kg)/(height in m)^2)
Collecte of Waist Circumference | at baseline
  Waist Circumference: measured in centimeters during routine care
Collecte of Body Composition | at baseline
  Body Composition (bioelectrical impedance analysis, BIA): when available, bioimpedance measures of fat mass and lean mass will be recorded))

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Hage, MD, PhD, Principal Investigator — Department of endocrinology, diabetology and nutrition, Ambroise Paré Hospital - A
Locations (1):
- Department of endocrinology, diabetology and nutrition, Ambroise Paré Hospital - APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No